CLINICAL TRIAL: NCT06722274
Title: Nutritional Habits Among People with and Without Diabetes in Upper Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Mohammed Ahmed Mohammed, resident doctor at internal medicine Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: Nutritional habits DM- Non DM
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: Nutritional habits
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: patients with diabetes
- Group B: healthy control (without diabetes)

SUMMARY:
Type2 Diabetes is a serious chronic disease associated with numerous complications. It is pandemic disease due to worsening of diatery habits and westernization of diet. These complications contribute to nearly half (46.1%) of deaths occurring in adults under 60, the working-age population. With this alarming increase, and in order to decrease complications and diabetes-related mortality, this health problem requires a comprehensive management plan where patients should be educated to make informed decisions about diet, exercise, weight, and medications, as recommended by the American Diabetes Association (ADA).

the aim of the study is -to detect nutritional habits in our locality among diabetic patients comparing to non diabetics.

DETAILED DESCRIPTION:
Recent analysis has reported that for the management of diabetes, only pharmacologic approaches are not sufficient. The management of diabetes is a multifactorial process involving life style and dietery factors that influence the treatment outcomes. There are also patient-related factors, such as self-care behaviors, that have a strong influence on glycemic intolerance.

Diabetes management necessitates both medication and lifestyle adjustments, which are associated with a decreased risk of death. people with T2DM find dietary advice confusing, contradictory, and report that understanding and making healthy eating choices are the most challenging parts of living with the condition. Therefore, national guidelines recommend that all patients with T2DM should receive individualized, ongoing dietary advice from a health professional with expertise in nutrition. The role standing of diet in controlling of diabetes is considered imperative; still, diabetes patients are unaware of how they should approach this issue to ensure good glycaemiccontrol .in Egypt no sufficient screening about diatery habits .hypothesis:there is difference in diatery habits between patients with and without diabetes

ELIGIBILITY:
Inclusion Criteria:

* adults participant whose age > 18or older .
* type 2 DM

Exclusion Criteria:

* Patients who have stroke patients who have dementia. CKD patients (as it affects appetite and diet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: diabetic cases from outpatient diabetic clinic, centre of diabetes and endocrine, Department of Internal medicine, Assiut university hospitals matched control
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
nutrition knowledge score | baseline
  nutrition knowledge score: the questionnaire consisted of three domains: knowledge, self-efficacy, and practice, with a total of 30 questions distributed as follows: 10 questions assessing knowledge, 7 questions assessing self-efficacy, and 13 questions assessing practice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bawazeer NM, Benajiba N, Alzaben AS. Translation, validity, and reliability of an Arabic version of the dietary questionnaire on nutrition knowledge, self-efficacy, and practice among Arab young adults. Asia Pac J Clin Nutr. 2023;32(2):196-205. doi: 10.6133/apjcn.202306_32(2).0002. PMID 37382317
- [Background] Sami W, Alabdulwahhab KM, Ab Hamid MR, Alasbali TA, Alwadani FA, Ahmad MS. Dietary Knowledge among Adults with Type 2 Diabetes-Kingdom of Saudi Arabia. Int J Environ Res Public Health. 2020 Jan 30;17(3):858. doi: 10.3390/ijerph17030858. PMID 32019083
- [Background] England CY, Thompson JL, Jago R, Cooper AR, Andrews RC. Development of a brief, reliable and valid diet assessment tool for impaired glucose tolerance and diabetes: the UK Diabetes and Diet Questionnaire. Public Health Nutr. 2017 Feb;20(2):191-199. doi: 10.1017/S1368980016002275. Epub 2016 Sep 9. PMID 27609314
- [Background] Patel YR, Gadiraju TV, Gaziano JM, Djousse L. Adherence to healthy lifestyle factors and risk of death in men with diabetes mellitus: The Physicians' Health Study. Clin Nutr. 2018 Feb;37(1):139-143. doi: 10.1016/j.clnu.2016.11.003. Epub 2016 Nov 11. PMID 27866759
- [Background] Saeedi P, Salpea P, Karuranga S, Petersohn I, Malanda B, Gregg EW, Unwin N, Wild SH, Williams R. Mortality attributable to diabetes in 20-79 years old adults, 2019 estimates: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2020 Apr;162:108086. doi: 10.1016/j.diabres.2020.108086. Epub 2020 Feb 15. PMID 32068099